CLINICAL TRIAL: NCT04621734
Title: Improving Retention of Nasoenteric Feeding Tubes in Pediatric Patients Using a Nasal Bridle
Brief Title: Retention of Nasoenteric Feeding Tubes in Pediatric Patients Using a Nasal Bridle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20190225H
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Feeding Tube Complication
MeSH Terms: interventions — Surgical Tape

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Nasal bridle to secure feeding tube (Active Comparator): The nasal bridle will be used to secure the nasoenteric feeding tube.
  Interventions: Device: AMT BridlePro Device
- Adhesive Tape use to secure feeding tube (Placebo Comparator): Adhesive tape will be used as standard of care to secure the nasoenteric feeding tube.
  Interventions: Device: Adhesive Tape

INTERVENTIONS:
Device: AMT BridlePro Device — A device used as an alternative securement method using the structure of the nasal cavity to secure the nasoenteric tube.
  Other Names: Applied Medical Technology (AMT) BridlePro Device
  Arms: Nasal bridle to secure feeding tube
Device: Adhesive Tape — Adhesive tape used to secure nasoenteric tube
  Other Names: Tape
  Arms: Adhesive Tape use to secure feeding tube

SUMMARY:
A study to compare tube dislodgment rates when a nasoenteric feeding tube is secured with adhesive tape vs the AMT BridlePro device.

DETAILED DESCRIPTION:
The adhesive tape will be the tape available in the unit and will be placed by the nurse or provider at the time of nasoenteric tube placement. The tape will be placed around the tube and secured to the cheek on the side of tube. The tape will be replaced as needed per nursing discretion when soiled or the adhesive properties are failing and this information will be tracked. The AMT BridlePro will be placed by the nurse or provider at the time of nasoenteric tube placement. Placement will use the BridlePro system included in the individual BridlePro packaging. Placement and securement will follow manufacturer recommendations and teaching. The BridlePro encircles the vomer bone of the nasal cavity to secure the tube. Sedation medication may be given per standard of care for nasoenteric tube placement at the discretion of the provider team but no separate or additional sedation medication will be given for securement with adhesive tape or the BridlePro.

ELIGIBILITY:
Inclusion Criteria:

* Need for nasoenteric feeding
* Admitted to University Hospital
* Age 0-18 years

Exclusion Criteria:

* Facial trauma
* Nasal airway obstructions
* Thrombocytopenia (<100 K/μL)
* s/p septoplasty
* Patients with vomer bone graft
* Nasoenteric feeding tube placed and secured prior to being screened for study
* Contraindication for the use of the BridlePro
* Does not meet inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Armijo, MD, Principal Investigator — University of Texas Health at San Antonio
Locations (1):
- University Health System, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Foster M, Armijo-Garcia V, Gelfond J, Meyer AD. Improving retention of pediatric feeding tubes with a nasal bridle: a randomized controlled trial. Trials. 2025 May 14;26(1):159. doi: 10.1186/s13063-025-08867-x. PMID 40369642

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Bridle to Secure Feeding Tube | Adhesive Tape Use to Secure Feeding Tube
Started | 17 | 18
Completed | 16 | 17
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Bridle to Secure Feeding Tube | Adhesive Tape Use to Secure Feeding Tube | Total
Number analyzed (Participants) | 17 | 18 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 18 | 35
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 6.5 [0.1 to 17.1] | 9.1 [0.1 to 17.7] | 7.8 [0.1 to 17.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 31
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Tube Dislodgements Per 10 Tube Days.
Description: The number of times the tube is dislodged for every 10 days of feeding tubes.
Time Frame: 10 days
Measure: Mean (Full Range); unit: Dislodgements
Arm/Group | Nasal Bridle to Secure Feeding Tube | Adhesive Tape Use to Secure Feeding Tube
Number analyzed (Participants) | 16 | 17
Dislodgements | 0.16 [0 to 10] | 2.11 [0 to 10]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Nasal Bridle to Secure Feeding Tube | Adhesive Tape Use to Secure Feeding Tube
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 1/17 | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nasal Bridle to Secure Feeding Tube (N=17) | Adhesive Tape Use to Secure Feeding Tube (N=18)
Skin Breakdown (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) — Skin breakdown at the site of the bridle or adhesive tape

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT04621734/Prot_SAP_000.pdf